CLINICAL TRIAL: NCT05114083
Title: Symptom Scoring for Predicting Vocal Cord Dysfunction (VCD)
Status: Withdrawn | Type: Observational
Why Stopped: personnel redeployment
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jonathan Parsons, Associate Professor of Internal Medicine, Ohio State University
Other Study IDs: 2014H0368
Record Dates: First submitted 2015-09-24; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Vocal Cord Dysfunction
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: symptom assessment — symptom assessment

SUMMARY:
Dr. Russell Traister, et al, describes a symptom scoring system based on retrospective chart review to help identify subjects with VCD. Dr. Traister assigned the following symptom scores: dysphonia (2), throat tightness (4), sensitivity to odors (3) and absence of wheezing (2). Patients scoring 4 or more points have a positive predictive value of 96% and a negative predictive value of 77% for VCD. This prospective study will look at a population of patients presenting to a large tertiary care referral center for symptoms of cough. Patients seen at the "Cough Clinic" are evaluated by a Pulmonologist and an Otolaryngologist. Each patient undergoes pulmonary function testing and VLS testing as part of the diagnostic workup. For this study the history would be expanded to include the 4 specific symptoms: dysphonia, throat tightness, sensitivity to odors and absence of wheezing. The symptoms will be scored and compared against the results of diagnostic testing to determine if these symptoms help predict those with vocal cord dysfunction (VCD).

DETAILED DESCRIPTION:
Vocal cord dysfunction (VCD) refers to the abnormal adduction of the vocal cords during breathing resulting in extrathoracic airway obstruction. These patients often complain of wheezing, cough and shortness of breath. Symptoms of VCD mimic asthma often leading to misdiagnosis and exposure to unneeded medications. Speech therapy rather than medications is the mainstay of treatment for VCD.

The gold standard diagnostic tool for detection of VCD is direct visualization of the vocal cords using flexible video assisted fiberoptic laryngoscopy (VLS). VCD is present if the cords constrict greater than 50% during the respiratory cycle. VLS is well tolerated however it is an invasive procedure and costly. Identifying patients who most likely have VCD for VLS testing would reduce health related expense and avoid unnecessary procedures. Dr. Russell Traister, et al, describes a symptom scoring system based on retrospective chart review to help identify subjects with VCD. Dr. Traister assigned the following symptom scores: dysphonia (2), throat tightness (4), sensitivity to odors (3) and absence of wheezing (2). Patients scoring 4 or more points have a positive predictive value of 96% and a negative predictive value of 77% for VCD.

This prospective study will look at a population of patients presenting to a large tertiary care referral center for symptoms of cough. Currently patients seen at the "Cough Clinic" are evaluated by a pulmonologist and an Otolaryngologist during their visit. Each patient undergoes pulmonary function testing and VLS testing as part of the diagnostic workup. For this study the history would be expanded to include the 4 specific symptoms described above and scores tabulated and compared against the results of diagnostic testing. The findings of this study will help providers understand the characteristics of patients with VCD and use this information when deciding which patients should be referred for VLS testing.

ELIGIBILITY:
Inclusion Criteria:

* All participants male and female,
* age 18 years and older
* presenting as new patients to the Cough Clinic

Exclusion Criteria:

* Participants less than 18 years of age and those attended by a guardian or an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants male and female, age 18 years and older presenting as new patients to the Cough Clinic will be asked to participate if they are not attended by a guardian or an interpreter. Everyone (regardless if they choose to participate or not) will receive current standard practice/care of the Cough Clinic for evaluation, testing and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Determine if symptom scoring can accurately predict vocal cord dysfunction | 1 year
  We will score each patient according to their symptoms of vocal cord dysfunction including; throat tightness (4 points), dysphonia (2 points), absence of wheezing (2 points), symptoms triggered by strong odors (3 points). A positive response will be assigned the score as indicated in parentheses behind each symptom. A negative response will be assigned zero points.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Parsons, MD, Principal Investigator — Ohio State University

REFERENCES:
- [Background] Parsons JP, Benninger C, Hawley MP, Philips G, Forrest LA, Mastronarde JG. Vocal cord dysfunction: beyond severe asthma. Respir Med. 2010 Apr;104(4):504-9. doi: 10.1016/j.rmed.2009.11.004. Epub 2009 Dec 4. PMID 19962874
- [Background] Wilson JJ, Theis SM, Wilson EM. Evaluation and management of vocal cord dysfunction in the athlete. Curr Sports Med Rep. 2009 Mar-Apr;8(2):65-70. doi: 10.1249/JSR.0b013e31819def3d. PMID 19276905
- [Background] Sterner JB, Morris MJ, Sill JM, Hayes JA. Inspiratory flow-volume curve evaluation for detecting upper airway disease. Respir Care. 2009 Apr;54(4):461-6. PMID 19327180
- [Background] Benninger C, Parsons JP, Mastronarde JG. Vocal cord dysfunction and asthma. Curr Opin Pulm Med. 2011 Jan;17(1):45-9. doi: 10.1097/MCP.0b013e32834130ee. PMID 21330824
- [Background] Traister RS, Fajt ML, Landsittel D, Petrov AA. A novel scoring system to distinguish vocal cord dysfunction from asthma. J Allergy Clin Immunol Pract. 2014 Jan-Feb;2(1):65-9. doi: 10.1016/j.jaip.2013.09.002. Epub 2013 Nov 2. PMID 24565771